CLINICAL TRIAL: NCT01929902
Title: Laparoscopic Aquamantys Device in General Surgery: A Prospective Observational Study to Evaluate the Efficacy and Accuracy
Brief Title: Evaluation of Efficacy and Accuracy of Aquamantys Device in General Surgery
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-13-04E
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2014-04

CONDITIONS: Cancer, Hepatocellular; Pancreatectomy
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Surgical Patients

SUMMARY:
The purpose of this study is to test the efficacy and accuracy of the Aquamantys device.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy of placement and accuracy of the Aquamantys device in 20 patients that require general surgery. High frequency electrosurgery is the application of frequency in the range of 300 kHz up to several MHz in order to coagulate or destroy tissue. Due to technological advancements, knowledge of how frequency and other physical modes interact with biological materials has become increasingly important in order for the surgeon to provide a safe and consistent surgery. The Aquamantys system utilizes radiofrequency energy and saline irrigation for cutting tissue and stopping excessive bleeding.

The Aquamantys system features the following:

1. Cone-shaped electrodes designed to aid blunt dissection;
2. Large bipolar electrode configuration allowing for hemostatic sealing across broad planes of tissue;
3. Bipolar electrodes alleviate the need for grounding pad;
4. Transcollation technology allows for controlled depth of energy penetration.

During surgery, the Aquamantys device will be utilized in order to stop excessive bleeding and to cut vessels. The patient will be monitored by the surgeon and research nurse coordinator before surgery, intra-operatively and post-operatively until discharge from the hospital. The study participant will follow-up post-operatively with the surgeon per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Indication for general surgery to include: liver resection and pancreatectomy
* Male or females age 18 years of age or older

Exclusion Criteria:

* Indication for emergency surgery
* Suspected inability, e.g. language problems or the inability to comply with trial procedures
* Employee at the investigational center, Sponsor or Sponsor's representative, relative or spouse of the investigator
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients age 18 years or older and in need of general surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Aquamantys Device | 1 year
  Efficacy of device will be measured based on intra-operative and post-operative complication variables: estimated blood loss, blood transfusion, complications intra-operative and post-operative.
Placement of Aquamantys Device | 1 year
  Evaluation of device placement will be measured based on vessel sealing variables: number of applications, vessel site, type of tissue to be sealed, number of failed and successful seals, tissue sticking, tissue color, thermal spread and desiccation.

SECONDARY OUTCOMES:
Device Complications | 1 year
  Functional evaluation of device based on the variable: device malfunction.

CONTACTS AND LOCATIONS:
Overall Officials: David Iannitti, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Healthcare System, Charlotte, North Carolina, United States